CLINICAL TRIAL: NCT06011135
Title: Exploring Worry in the Context of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS): A Qualitative Study
Brief Title: Exploring Worry in CFS/ME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 320892
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention - qualitative study only using semi-structured interview

SUMMARY:
This study will be building on the findings of Kalfas et al 2022 paper exploring the prevalence of generalised worry in patients with Myalgic Encephalomyelitis/ Chronic Fatigue Syndrome (ME/CFS) before and after Cognitive Behavioural Therapy (CBT). The research was conducted in South London and Maudsley NHS Foundation Trust's (SLaM) Persistent Physical Symptoms Research and Treatment Unit. Previous research has indicated a bidirectional relationship between fatigue and worry (Kalfas et al., 2022); the findings of this paper suggest both that many ME/CFS patients experience comorbid problematic generalised worry and that there is a positive association between severity of worry and levels of fatigue (Kalfas et al, 2022). It appears that CBT for ME/CFS indirectly treats worry, however effect sizes are small to moderate, and treatment outcomes may improve if CBT treatments incorporate strategies that target generalised worry (Kalfas et al 2022). The aims of this project are to further explore worry in this group of patients through qualitative methods.

DETAILED DESCRIPTION:
A recent study carried out in SLaM explored how common worry is in people who have received Cognitive Behavioural Therapy (CBT) for CFS/ME. Over 70% were struggling with worry, and the more severe their level of worry was, the more severe their fatigue was likely to be. Indirectly, CBT appeared to slightly reduce how much people struggle with worry which queried: could CBT for CFS/ME be improved if we had a better understanding of worry in this context?

Worry in CFS/ME is not well understood; the present study aims to explore worry in people who have a diagnosis of CFS/ME through qualitative interviews, with the hope of gathering information to inform future treatments.

CFS/ME is a long-term condition, meaning treatments aim to manage rather than cure. It can range from a mild illness to severely disabling. National UK guidance states CBT should be offered to those living with CFS/ME. CBT treatments recognise that how our bodies function is closely linked to our thoughts, feelings, and behaviour. Research into CBT for CFS/ME shows it can improve levels of fatigue, distress, and how much people can do physically, however, in most studies improvements are small. CBT has stronger evidence for treating mental health difficulties, such as anxiety and depression. These difficulties are more common in people who have a diagnosis of CFS/ME, particularly Generalised Anxiety Disorder (GAD) which has been reported to be as high as 34%, in comparison to up to 7% of the general population. There has been little research into anxiety and how it affects fatigue, but research has identified a 'bidirectional relationship' between the two. This study is building on the finding that over 70% of people with CFS/ME could be struggling with significant worry that doesn't meet the criteria for GAD but causes distress and impacts fatigue.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of ME/CFS according to NICE criteria;
* have agreed to CBT for ME/CFS following their initial assessment;
* are/were struggling with comorbid generalised worry as determined by a score of 45 or above on the Penn State Worry Questionnaire (collected routinely with all patients referred to the service).
* Informed consent to taking part in the study

Exclusion Criteria:

* Patients who have been closed to the service longer than 3 months
* Patients with a diagnosis of long-Covid
* Patients who are under 18
* Patients who do not have a diagnosis of CFS/ME
* Patients who have not agreed to CBT for CFS/ME as part of their treatment
* Patients who score below the threshold on the PSWQ

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A purposeful sample of patients will be recruited from SLaM's Persistent Physical Symptoms Research and Treatment Unit. We are interested to collect the views of patients pre, during, and post CBT treatment to support with the secondary aim of the project which is to use the discussions to make recommendations for targeted CBT treatments. Patients will therefore be eligible to participate at any stage of their treatment following initial assessment.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Exploration of how people with a diagnosis of CFS/ME experience worry | 31/05/2024
How can this exploration of how people with a diagnosis of CFS/ME experience worry inform future research into targeted CBT interventions in the context of ME/CFS. | 31/05/2024

CONTACTS AND LOCATIONS:
Locations (1):
- Kings College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data to be shared with other researchers.